CLINICAL TRIAL: NCT03160794
Title: Phase II Study: [18F]DCFPyL PET/MRI for Personalizing Prostate Cancer Subclinical Metastatic Ablative MR-guided Radiotherapy (MRgRT)
Brief Title: Prostate Cancer Subclinical Metastatic Ablative MR-guided Radiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-5532
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Post Prostatectomy
Keywords: Prostate cancer; stereotactic ablative radiotherpy; PET/MR
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18F] DCFPyL PET/MRI (Experimental): [18F] DCFPyL PET/MRI scans for patients with recurrent disease after radical prostatectomy and adjuvant/salvage radiotherapy.
  Lesions identified through [18F] DCFPyL PET/MRI will be treated with stereotactic ablative radiotherapy (SABR) or surgery.
  Interventions: Diagnostic Test: [18F]DCFPyL PET/MRI scan; Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Diagnostic Test: [18F]DCFPyL PET/MRI scan — PET/MRI imaging using the radiotracer, [18F]DCFPyL
Radiation: Stereotactic Ablative Radiotherapy — SABR as treatment for lesions identified using [18F]DCFPyL PET/MRI

SUMMARY:
In the clinical scenario of recurrent prostate cancer (PCa) post local therapy, current standard studies (bone scan and computed tomography) commonly fail to identify the recurrent disease location. In this study the investigator aims to prospectively map recurrent disease with the unique combination of whole-body MR anatomical imaging combined with a new high-sensitivity and PCa-specific PET probe (PSMA-targeted: [18F]DCFPyL) to provide precise localization information to target disseminated tumor deposits in men presenting with rising PSA after prostatectomy and radiotherapy (maximal local therapies). Moreover, we will consequently treat all identified disease with image-guided stereotactic ablative radiotherapy (SABR), which has shown tantalizing results achieving excellent tumor eradication rates with minimal toxicities. This study is uniquely positioned to enable the discovery of new biomarkers and the correlation of prognostic tests (e.g. genomic signatures) from the initial prostatectomy specimen with the PET-MR/CT imaging results and curative-intent treatment outcomes.

The significance of the proposed work towards a measurable impact in PCa care is important to emphasize. The study team believes this novel curative-intent approach will transform lives, as opposed to therapies that transiently impact incurable disease stages. Herein, the focus is on patients at the earliest point of the disease spectrum of recurrent PCa after curative-intent treatments. Our hypothesis is that PSMA-targeted [18F]DCFPyL PET-MR/CT allows earlier detection and localization of defined metastatic targets in these patients, at a stage amenable to image-guided curative-intent therapy.

ELIGIBILITY:
* ECOG performance status of 0-2
* Absence of significant comorbidities rendering patient nor suitable for curative ablative approaches
* No history of non-skin malignancy
* Histological evidence of prostate adenocarcinoma on previous radical prostatectomy.
* No use of any form of hormonal therapy in the previous 12 months, or intention to start HT at time of enrollment.
* Normal serum testosterone level ascertained within 4-6 weeks of enrollment
* Absence of known metastatic disease
* Radiological studies without evidence of regional or distant metastases: CT abdomen-pelvis and bone scan within previous 3 months
* Able to lie supine at least 60 minutes to comply with imaging and treatment.
* Absence of impaired renal function (calculated GFR > 30mL/min)
* Absence of sickle cell disease or other hemoglobinopathies
* No other medical conditions deemed by the PI to make patient ineligible for PET/MR scanning or SABR

No contraindications to MRI:

* Subject must weigh <136kg (scanner weight limit)
* Subject must not have pacemakers, cerebral aneurysm clips, shrapnel injury, or implantable electronic devices not compatible with MRI
* Prior anaphylactic reaction to gadolinium

Rising PSA after maximal local therapies (radical prostatectomy and either adjuvant or salvage radiotherapy):

* Three documented PSA rises, at least 1 month apart from post radiotherapy.
* PSA value >0.1 and < 3 ng/mL, within 4-6 weeks of enrollment
* No use of any forms of ADT in the previous 12 months nor contemplated to be used at time of study enrollment. Salvage ADT to be started when PSA reaches a value of 6.0ng/ml or greater.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-23 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To determine if [18F]DCFPyL PET-MR/CT can identify early oligometastatic disease in patients with a rising PSA and negative staging (CS and BS) after standard-of-care maximal local therapies. | 3 years
  Endpoint: Detection rates and performance metrics of [18F]DCFPyL PET-MR/CT in the post-prostatectomy plus adjuvant/salvage RT setting.
To determine if treating PET-MR/CT identified lesions with curative-intent treatment (e.g. stereotactic body radiation therapy or surgery) associated with favorable preliminary measures of clinical performance. | 3 Years
  * Proportion of patients achieving biochemical response: detectable PSA (<0.05ng/mL) in 2 consecutive measurements (at least 2 weeks apart) within 6 months of treatment); or > 50% PSA decline in 2 separate measurements at least 1 month apart within 6 months of treatment
  * Metabolic [18F]DCFPyL response rate after treatment
  * Treatment-related toxicities incidence as defined by CTCAE v4.0
  * Time to initiation of salvage ADT after treatment

SECONDARY OUTCOMES:
Correlation between PSA kinetics and PET imaging parameters | 6 months post SABR
  To explore the correlation between PSA kinetics and PET imaging parameters (SUV, dynamic data, volumetric studies)
Correlate between tissue biomarker and distant disease | 3 years
  To explore the correlation between tissue biomarkers from prostatectomy specimen (e.g. genomic signatures) and [18F]DCFPyL PET/MR-detected distant disease

OTHER OUTCOMES:
[18F]DCFPyL PET/MR and PET/CT comparison | 3 years
  To determine concordance and compare performance between [18F]DCFPyL PET/MR and PET/CT
Concordance of PET-MR/CT finding and histological confirmation of metastatic foci. | 3 years
  To determine the concordance of PET-MR/CT findings and histological confirmation of metastatic foci.
Biomarker correlates | 3 years
  To explore blood, urine and tissue biomarker correlates of imaging features and radiotherapy tumour resposnse.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Berlin, MD, Principal Investigator — Princess Margaret Cancer Centre - University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Glicksman RM, Metser U, Valliant J, Chung PW, Fleshner NE, Bristow RG, Green D, Finelli A, Hamilton R, Stanescu T, Hussey D, Catton C, Gospodarowicz M, Warde P, Bayley A, Breen S, Vines D, Jaffray DA, Berlin A. [18F]DCFPyL PET-MRI/CT for unveiling a molecularly defined oligorecurrent prostate cancer state amenable for curative-intent ablative therapy: study protocol for a phase II trial. BMJ Open. 2020 Apr 22;10(4):e035959. doi: 10.1136/bmjopen-2019-035959. PMID 32327479